CLINICAL TRIAL: NCT04793529
Title: Is Involucrin Has a Role in Verruca Vulgaris? A Clinical and Immunohistochemical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Essam Mohamed El-sayed Akl, Assistant Professor, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC-2-3-2021
Record Dates: First submitted 2021-03-04; First posted 2021-03-11 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Verruca Vulgaris; Involucrin
MeSH Terms: conditions — Warts | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cholecalciferol injection (Experimental)
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — Cholecalciferol injection

SUMMARY:
Vitamin D3 plays important role in keratinocyte differentiation and had been used recently in verruca vulgaris. Aim of the work: To assess the expression of involucrin in verrucae vulgaris before and after injection of vitamin D3. Subjects and Methods: This study included 60 patients with verrucae vulgaris subjected to intralesional injection of vitamin D3 at three weeks interval for a maximum of five sessions. Immunohistochemical assessment of involucrin was done before and after injection and compared to skin biopsies from 30 healthy individuals

ELIGIBILITY:
Inclusion criteria:

Patients with multiple verruca vulgaris Patients with with verrucae vulgaris with size more than 3 cm

Exclusion Criteria:

Patients with a past history of allergic response to vitamin D. Pregnant or lactating females. Hepatic patients. Renal patients. Patients with bleeding tendency.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Resolution of verrucae | 3 months
  Decrease of verrucae size Decrease of verrucae number

SECONDARY OUTCOMES:
Involucrin expression | 3 months
  Change of expression pattern of involucrin by immunohistochemical study Change of expression grade of involucrin by immunohistochemical study

CONTACTS AND LOCATIONS:
Locations (1):
- Essam Mohamed El-sayed Akl, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: Undecided